CLINICAL TRIAL: NCT00141778
Title: RAAS, Inflammation, and Post-operative AF
Brief Title: Renin-angiotensin-aldosterone System (RAAS), Inflammation, and Post-Operative Atrial Fibrillation (AF)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy J. Brown, Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 040385; R01HL077389 (NIH); NCT00134862 (obsolete NCT alias)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ramipril; Angiotensin-Converting Enzyme Inhibitors; Spironolactone; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): matched placebo pills daily beginning 4-7 days before surgery and continuing through discharge
  Interventions: Drug: Placebo
- Ramipril (Experimental): Ramipril daily (2.5mg, increased to 5mg) beginning 4 to 7 days before surgery and continuing through discharge
  Interventions: Drug: Ramipril
- Spironolactone (Experimental): Spironolactone 25mg daily beginning 4 to 7 days before surgery and continuing through discharge
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Placebo — Matching placebo taken once a day
  Other Names: Placebo tablet
  Arms: Placebo
Drug: Ramipril — Taken orally, once a day
  Other Names: Angiotensin-converting enzyme inhibitor
  Arms: Ramipril
Drug: Spironolactone — Taken orally, once a day
  Other Names: Mineralocorticoid Receptor Antagonist
  Arms: Spironolactone

SUMMARY:
Atrial fibrillation (AF) is the most prevalent, sustained type of irregular heartbeat and affects over 2 million Americans. Post-operative AF, which leads to significant morbidity and a prolonged hospital stay, complicates 20% to 40% of cardiopulmonary bypass (CPB) surgical procedures. While recent studies indicate that interruption of the renin-angiotensin-aldosterone system by either angiotensin-converting enzyme (ACE) inhibition or AT1 receptor antagonism decreases the incidence of AF following a heart attack or cardioversion (electric shock to the heart), its effect on the incidence of post-operative AF has not been throughly studied. Studies in both animals and humans suggest that inflammation-induced atrial remodeling plays an important role in the cause of AF. Recent studies also provide evidence that activation of the renin-angiotensin-aldosterone system induces inflammation, myocyte injury, proarrhythmic electrical remodeling, and fibrosis through aldosterone.

DETAILED DESCRIPTION:
AF is the most prevalent, sustained type of irregular heartbeat and affects over 2 million Americans. Post-operative atrial fibrillation(AF), which leads to significant morbidity and a prolonged hospital stay, complicates 20% to 40% of CPB surgical procedures. While recent studies indicate that interruption of the renin-angiotensin-aldosterone system by either angiotensin-converting enzyme(ACE) inhibition or angiotensin II subtype 1 (AT1) receptor antagonism decreases the incidence of AF following a heart attack or cardioversion (electric shock to the heart), its effect on the incidence of post-operative AF has not been throughly studied. Studies in both animals and humans suggest that inflammation-induced atrial remodeling plays an important role in the cause of AF. Recent studies also provide evidence that activation of the renin-angiotensin-aldosterone system induces inflammation, myocyte injury, proarrhythmic electrical remodeling, and fibrosis through aldosterone.

This study will evaluate the effectiveness of ACE inhibition and aldosterone receptor antagonism at decreasing inflammation and AF following cardiopulmonary bypass (CPB) surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective valvular heart surgery, coronary artery bypass grafting
2. If female, must be postmenopausal for at least 1 year, status-post surgical sterilization, or if of childbearing potential, utilizing adequate birth control and willing to undergo urine beta-hcg testing prior to drug treatment and throughout the study

Exclusion Criteria

1. History of AF other than remote paroxysmal AF
2. Ejection fraction less than 30%
3. Evidence of coagulopathy (INR greater than 1.7 without warfarin therapy)
4. Emergency surgery
5. History of ACE inhibitor-induced angioedema
6. Low blood pressure (systolic blood pressure less than 100 mmHg and evidence of hypoperfusion)
7. Hyperkalemia (potassium level greater than 5.0 milliequivalents (mEq)/L at study entry)
8. Impaired kidney function (serum creatinine level greater than 1.6 mg/dl)
9. Any underlying or acute disease requiring regular medication that could possibly cause complications or make implementation of the study or interpretation of the study results difficult
10. Inability to discontinue current ACE inhibitor, AT1 receptor antagonist, or aldosterone receptor antagonist therapy
11. History of alcohol or drug abuse
12. Treatment with any investigational drug in the month prior to study entry
13. Mental condition that makes it impossible to understand the nature, scope and possible consequences of the study
14. Inability to comply with the study procedures (e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study)
15. Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2005-04; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Brown, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Billings FT 4th, Pretorius M, Siew ED, Yu C, Brown NJ. Early postoperative statin therapy is associated with a lower incidence of acute kidney injury after cardiac surgery. J Cardiothorac Vasc Anesth. 2010 Dec;24(6):913-20. doi: 10.1053/j.jvca.2010.03.024. PMID 20599398
- [Result] Fleming GA, Murray KT, Yu C, Byrne JG, Greelish JP, Petracek MR, Hoff SJ, Ball SK, Brown NJ, Pretorius M. Milrinone use is associated with postoperative atrial fibrillation after cardiac surgery. Circulation. 2008 Oct 14;118(16):1619-25. doi: 10.1161/CIRCULATIONAHA.108.790162. Epub 2008 Sep 29. PMID 18824641
- [Result] Pretorius M, Murray KT, Yu C, Byrne JG, Billings FT 4th, Petracek MR, Greelish JP, Hoff SJ, Ball SK, Mishra V, Body SC, Brown NJ. Angiotensin-converting enzyme inhibition or mineralocorticoid receptor blockade do not affect prevalence of atrial fibrillation in patients undergoing cardiac surgery. Crit Care Med. 2012 Oct;40(10):2805-12. doi: 10.1097/CCM.0b013e31825b8be2. PMID 22824930
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Sidorova TN, Mace LC, Wells KS, Yermalitskaya LV, Su PF, Shyr Y, Atkinson JB, Fogo AB, Prinsen JK, Byrne JG, Petracek MR, Greelish JP, Hoff SJ, Ball SK, Glabe CG, Brown NJ, Barnett JV, Murray KT. Hypertension is associated with preamyloid oligomers in human atrium: a missing link in atrial pathophysiology? J Am Heart Assoc. 2014 Dec 2;3(6):e001384. doi: 10.1161/JAHA.114.001384. PMID 25468655
- [Derived] Billings FT 4th, Pretorius M, Schildcrout JS, Mercaldo ND, Byrne JG, Ikizler TA, Brown NJ. Obesity and oxidative stress predict AKI after cardiac surgery. J Am Soc Nephrol. 2012 Jul;23(7):1221-8. doi: 10.1681/ASN.2011090940. Epub 2012 May 24. PMID 22626819

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 2005 and 2010 from Vanderbilt University Medical Center and Brigham and Women's Hospital
Pre-assignment Details: One week to four days prior to surgery, patients were randomized to treatment with placebo, ramipril or spironolactone. Preexisting ACE inhibitor, angiotensin receptor blocker, or MR antagonist use was stopped at randomization. Four hundred and fifty-eight patients met inclusion and were randomized
Groups:
- Placebo: Placebo Group
- Ramipril: Angiotensin-Converting Enzyme Inhibitor Group. Ramipril was given as 2.5 mg the first 3 days followed by 5 mg/day, with the dose reduced to 2.5 mg/day on the first postoperative day only.
- Spironolactone: Mineralocorticoid Receptor (MR) Antagonist Group.Spironolactone was given as 25 mg/day.
Period: Randomization Prior to Study Med
Arm/Group | Placebo | Ramipril | Spironolactone
Started | 152 | 153 | 153
Completed | 147 | 151 | 147
Not Completed | 5 | 2 | 6
Not completed — Withdrawal by Subject | 5 | 2 | 6
Period: Started Study Medication
Arm/Group | Placebo | Ramipril | Spironolactone
Started | 147 | 151 | 147
Completed | 145 | 144 | 143
Not Completed | 2 | 7 | 4
Not completed — Met safety criteria for discontinuation | 2 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Difficulty Swallowing | 0 | 1 | 0
Not completed — Chest Discomfort | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ramipril: Angiotensin-converting enzyme inhibitor group
- Spironolactone: Mineralocorticoid Receptor (MR) Antagonist group
- Total: Total of all reporting groups
Arm/Group | Placebo | Ramipril | Spironolactone | Total
Number analyzed (Participants) | 147 | 151 | 147 | 445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 94 | 101 | 99 | 294
  >=65 years | 53 | 50 | 48 | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 60.0 (12.0) | 58.7 (12.3) | 59.2 (12.3) | 59.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 45 | 51 | 149
  Male | 94 | 106 | 96 | 296
Region of Enrollment [Number; unit: participants]
  United States | 147 | 151 | 147 | 445

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Atrial Fibrillation
Description: The primary endpoint of the study was the percentage of patients with electrocardiographically confirmed AF of at least 10 secs duration at any time following the end of surgery until hospital discharge, an average from 5.7 days in the ramipril group to 6.8 days in the placebo group. Patients were monitored continuously on telemetry throughout the postoperative period until discharge. Electrocardiograms were obtained for any rhythm changes detected on telemetry monitoring, and in addition, electrocardiograms were performed preoperatively, at admission to the intensive care unit, and daily starting on postoperative day 1. All electrocardiograms and rhythm strips were reviewed in a blinded fashion by a single cardiac electrophysiologist.
Time Frame: Measured from admission to the ICU until discharge from hospital
Population: Four hundred fifty-eight patients were randomized. Of these 445 took study medication and were included in the intention-to-treat analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
percentage of patients | 27.2 | 27.8 | 25.9
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Discrete variables were compared among treatment groups with a chi-square test; Test type: Superiority or Other; p = 0.95, Chi-squared

2. Secondary Outcome: Acute Renal Failure
Description: Percentage of patients with a creatinine concentrations >2.5mg/dl
Time Frame: Measured until the time of hospital discharge, from 5.7 to 6.8 days on average, depending on the study group.
Population: The intention-to-treat analysis included anyone who had received any study medication.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
percentage of patients | 5.4 | 0.7 | 0.7
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Test type: Superiority or Other; p = 0.006, Chi-squared

3. Secondary Outcome: Hypotension
Description: Percentage of patients with hypotension defined as a systolic blood pressure <90 mmHg and/or prolonged requirement for vasopressor use.
Time Frame: Measured during and after surgery, until discharge, from 5.7 to 6.8 days on average.
Population: The intention-to-treat analysis included anyone who had received any medication.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
percentage of patients | 5.4 | 10.6 | 10.2
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Test type: Superiority or Other; p = 0.15, Chi-squared

4. Secondary Outcome: Hypokalemia
Description: Percentage of patients who had a serum potassium concentrations <3.5 milliequivalents (mEq)/L
Time Frame: Measured until the time of hospital discharge, which was an average of 5.7 to 6.8 days depending on the treatment arm.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
percentage of patients | 11.6 | 13.8 | 6.8
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Test type: Superiority or Other; p = 0.14, Chi-squared

5. Secondary Outcome: Time to Tracheal Extubation
Description: It is the time in minutes that it took to extubate the patient after surgery.
Time Frame: It is the time (in minutes) from admission to the ICU until tracheal extubation
Population: The intention-to-treat analysis included all patients who received any study medication.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
minutes | 1091.3 (3067.3) | 970.1 (3548.1) | 576.4 (761.5)
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Test type: Superiority or Other; p = 0.56, Kruskal-Wallis

6. Secondary Outcome: Length of Hospital Stay (Days)
Time Frame: Measured from the day of surgery until the time of hospital discharge
Population: The intention-to-treat analysis included anyone who had received any study medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
days | 6.8 (8.2) | 5.7 (3.2) | 5.8 (3.4)
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Test type: Superiority or Other; p = 0.15, Kruskal-Wallis

7. Secondary Outcome: Death
Description: The percentage of patients in each study arm who died.
Time Frame: Measured until the time of hospital discharge
Population: The intention-to-treat analysis included all patients who received any study medication.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
percentage of patients | 1.4 | 2.0 | 0
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Test type: Superiority or Other; p = 0.38, Chi-squared

8. Secondary Outcome: Stroke
Description: Percentage of patients in each study group who experience a cerebrovascular event, confirmed by CT.
Time Frame: Measured until the time of hospital discharge, from 5.7 to 6.8 days on average depending on the study arm.
Population: The intention-to-treat analysis included all those who received any study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 147 | 151 | 147
percentage of patients | 2.7 | 1.3 | 2.0
Statistical Analysis 1: Comparison: Placebo vs Ramipril vs Spironolactone; Test type: Superiority or Other; p = 0.65, Chi-squared

9. Secondary Outcome: Perioperative Interleukin(IL)-6 Concentrations
Description: Interleukin-6 was measured at several time points (see time points in table) over the course of the study
Time Frame: Perioperative period
Population: All participants included in the intention-to-treat analysis who had available plasma samples.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 136 | 136 | 140
pg/ml
  Initiation of surgery | 4.7 (6.7) | 4.6 (7.1) | 6.6 (10.2)
  30min intraop | 12.0 (18.4) | 20.5 (72.6) | 11.3 (20.2)
  60min intraop | 15.6 (20.1) | 28.8 (100.9) | 17.4 (29.4)
  Postop | 130.0 (213.7) | 202.1 (668.7) | 145.7 (427.1)
  Postoperative day 1 | 119.0 (143.1) | 171.0 (208.6) | 164.9 (200.2)
  Postoperative day 2 | 100.3 (106.8) | 95.5 (90.8) | 109.6 (116.9)

10. Secondary Outcome: Perioperative Plasminogen Activator Inhibitor-1 (PAI-1) Concentrations
Description: Plasminogen activator inhibitor-1 (PAI-1) was measured at several time points (see table) over the course of the study.
Time Frame: Perioperative period
Population: PAI-1 was measured in all subjects in the intention-to-treat analysis for which plasma was available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 135 | 133 | 136
ng/mL
  Initiation of surgery | 19.6 (16.6) | 16.2 (11.9) | 17.3 (12.0)
  30min intraop | 19.2 (10.7) | 19.7 (12.5) | 17.3 (10.9)
  60min intraop | 21.0 (10.9) | 22.0 (13.7) | 20.1 (11.7)
  Postop | 36.4 (24.6) | 38.9 (28.0) | 34.0 (22.3)
  Postoperative day 1 | 55.2 (43.8) | 47.9 (31.4) | 48.9 (35.0)
  Postoperative day 2 | 28.1 (20.4) | 25.7 (17.9) | 31.0 (30.5)

11. Secondary Outcome: Perioperative C-reactive Protein (CRP) Concentrations
Description: C-reactive protein was measured at several time points (see table) over the course of the study.
Time Frame: Perioperative period
Population: CRP was measured in all subjects from the intention-to-treat analysis for which plasma was available at those time points.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | Ramipril | Spironolactone
Number analyzed (Participants) | 127 | 129 | 126
ug/mL
  Initiation of surgery | 4.1 (6.8) | 4.3 (10.8) | 3.9 (7.3)
  Postoperative day 1 | 51.4 (40.0) | 49.9 (38.5) | 64.3 (115)
  Postoperative day 2 | 134.8 (137.4) | 131.0 (281.5) | 127.8 (84.8)
  Postoperative day 3 | 128.3 (88.7) | 164.8 (416.5) | 189.4 (476.0)
  Postoperative day 4 | 94.1 (67.3) | 105.2 (96.6) | 126.5 (95.4)

ADVERSE EVENTS:
Time Frame: Duration of hospital stay, which averaged from 5.7 to 6.8 days depending on the study arm.
Description: The intention-to-treat analysis included all subjects who received any study drug.
Arm/Group | Placebo | Ramipril | Spironolactone
Serious Adverse Events (participants affected / at risk) | 8/147 | 6/151 | 5/147
Other Adverse Events (participants affected / at risk) | 17/147 | 21/151 | 15/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=147) | Ramipril (N=151) | Spironolactone (N=147)
Death (General disorders) | 2 (2) | 3 (3) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 8 (8) | 1 (1) | 1 (1) — Creatinine >2.5mg/dL
Stroke (Nervous system disorders) | 4 (4) | 2 (2) | 3 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=147) | Ramipril (N=151) | Spironolactone (N=147)
Hypotension (Cardiac disorders) | 8 (8) | 16 (16) | 15 (15)
Hypokalemia (General disorders) | 17 (17) | 21 (21) | 10 (10) — Potassium <3.5 milliequivalents (mEq)/L postoperative day 1-4
Hyperkalemia (General disorders) | 1 (1) | 1 (1) | 1 (1) — Potassium >5.5 milliequivalents (mEq)/L

LIMITATIONS AND CAVEATS:
We excluded patients with an ejection fraction less than 30% or a creatinine above 1.6 and therefore the results are not applicable to patients with left ventricular dysfunction or more severe chronic kidney disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No